CLINICAL TRIAL: NCT03505749
Title: A Trauma Informed Adaptation of Mindfulness-Based Relapse Prevention for Women in Substance Use Treatment: A Randomized-controlled Pilot Trial
Brief Title: A Trauma Informed Adaptation of Mindfulness-Based Relapse Prevention for Women in Substance Use Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific University (Other)
Responsible Party: Principal Investigator, Vanessa Somohano, Graduate Student, Pacific University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R36DA043554-01A1 (NIH)
Record Dates: First submitted 2018-04-07; First posted 2018-04-23 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Substance Use Disorders; Post Traumatic Stress Disorder
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were made unaware of whether they were being randomized to the treatment or control group condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TI-MBRP (Experimental): Trauma Informed-Mindfulness-Based Relapse Prevention (TI-MBRP) will be a 4-week intervention integrating trauma intervention approaches based on Cognitive Processing Therapy (CPT) into standard Mindfulness-Based Relapse Prevention (MBRP). TI-MBRP honors the spirit and cognitive-behavioral foundation of MBRP while introducing components of CPT. Each TI-MBRP session will include mindfulness practices that bring awareness to cognitive and behavioral processes of substance abuse, and how substance use may function as a mechanism to cope with trauma symptoms. Clients are trained to observe internal, triggering stimuli without reactively attempting to avoid these experiences through substance use as well as complete exercises that promote cognitive and emotional processing of traumatic events.
  Interventions: Behavioral: Trauma Informed Mindfulness-Based Relapse Prevention
- Standard MBRP (Active Comparator): The Treatment as Usual (TAU) group implemented for this trial will be the standard protocol for Mindfulness-Based Relapse Prevention (MBRP). MBRP is a 4-week exposure-based intervention that integrates integrating mindfulness and acceptance-based techniques with cognitive-behavioral approaches and psycho-education to increase awareness of patterns associated with addictive behaviors and individual factors precipitating and maintaining substance use. These skills are also used to train individuals in responding skillfully in high-risk situations associated with use.
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Trauma Informed Mindfulness-Based Relapse Prevention — Trauma Informed-Mindfulness-Based Relapse Prevention (TI-MBRP) will be a 4-week intervention integrating trauma intervention approaches based on Cognitive Processing Therapy (CPT) into standard Mindfulness-Based Relapse Prevention (MBRP). TI-MBRP honors the spirit and cognitive-behavioral foundation of MBRP while introducing components of CPT. Each TI-MBRP session will include mindfulness practices that bring awareness to cognitive and behavioral processes of substance abuse, and how substance use may function as a mechanism to cope with trauma symptoms. Clients are trained to observe internal, triggering stimuli without reactively attempting to avoid these experiences through substance use as well as complete exercises that promote cognitive and emotional processing of traumatic events.
  Other Names: TI-MBRP
  Arms: TI-MBRP
Behavioral: Treatment As Usual (TAU) — The Treatment as Usual (TAU) group implemented for this trial will be the standard protocol for Mindfulness-Based Relapse Prevention (MBRP). MBRP is a 4-week exposure-based intervention that integrates integrating mindfulness and acceptance-based techniques with cognitive-behavioral approaches and psycho-education to increase awareness of patterns associated with addictive behaviors and individual factors precipitating and maintaining substance use. These skills are also used to train individuals in responding skillfully in high-risk situations associated with use.
  Other Names: Mindfulness-Based Relapse Prevention (MBRP)
  Arms: Standard MBRP

SUMMARY:
More than 90% of women in substance use treatment report history of physical and/or sexual trauma, and up to 60% meet criteria for both substance use disorder (SUD) and Post Traumatic Stress Disorder (PTSD). PTSD typically precedes onset of SUD, with substances used as a means to cope with physiological, psychological, and emotional symptoms resulting from the trauma. Women with PTSD experience greater severity of addiction symptoms, readmit into treatment more frequently than women without PTSD, and tend to have poorer treatment outcomes. Due to increased risk for exacerbation of PTSD on SUD severity and treatment success, and the specific vulnerabilities and needs of women with this comorbidity, SUD treatments that target both substance use and trauma recovery are needed. However, few interventions target both SUD and PTSD concurrently, and fewer still are specific to women.

Mindfulness-Based Relapse Prevention (MBRP) has been shown to decrease craving, relapse rates, and quantity/frequency of use across several substances, and has shown acceptability in diverse populations. MBRP integrates mindfulness practices with cognitive behavioral and exposure-based approaches to increase self-regulatory skills while experiencing triggers previously associated with substance use, including challenging affective states such as those common to experienced trauma. Adapting MBRP to incorporate trauma education and treatment approaches has the potential to effectively treat women with the dual vulnerabilities of trauma history and SUD.

The current study is thus designed to determine feasibility, acceptability, and initial efficacy of an adapted Trauma-Informed Mindfulness-Based Relapse Prevention (TI-MBRP) intervention for women in substance use treatment settings who have PTSD. TI-MBRP integrates trauma education and treatment approaches drawn from Cognitive Processing Therapy (CPT) into the standard MBRP protocol to provide a trauma-informed approach to treating women in substance use treatment settings. The current proposal will evaluate TI-MBRP, using a randomized, pre-post design, with 100 women in residential substance abuse treatment. Participants will be randomly assigned to participate in a 4-week TI-MBRP intervention or to continue with treatment as usual (TAU). Assessments will be collected pretest, posttest, and at one-month follow-up. Data from this study will lay the groundwork for a larger scale clinical trial to determine the efficacy of TI-MBRP.

DETAILED DESCRIPTION:
Approximately 4.7 million women in the US experience sexual and/or physical interpersonal violence (IPV) each year, and 46% experience IPV in their lifetime. More than 50% of interpersonal related violence occurs before age 25. In addition to acute, chronic and fatal injuries caused by IPV, women survivors of trauma (WST) are also at greater risk for organ and immune system diseases due to chronic stress, reproductive dysfunctions and complications during pregnancy, psychological disorders, and the inability to access health care services and social support. Estimated medical and mental health care costs for WST are $8.3 billion dollars per year, as well as $8 million dollars lost in paid workdays. Additionally, annual health care cost of survivors can persist up to 15 years after the cessation of abuse.

More than 90% of women admitted into substance use treatment settings have experienced IPV, and 30-60% meet criteria for comorbid SUD and PTSD. IPV typically precedes the onset of substance abuse as a means to cope with intense physiological, psychological, and emotional symptoms attributed to the event. Research has demonstrated that for women, PTSD symptoms may mediate the relationship between IPV and problematic SU. Women with PTSD symptoms and SUD also experience greater severity of addiction symptoms compared to men, and often readmit into treatment more frequently than men or women without traumatic histories. Evidence also suggests that PTSD symptoms and SU yields poorer treatment outcomes than any other comorbid disorder, or than SUD or PTSD alone. Due to these high rates of comorbidity and interrelationship of symptoms, particularly in women, integrated treatments targeting both substance use and trauma recovery are needed. However, few such evidence-based interventions (EBIs) are available for WST in substance use treatment settings. The few EBIs addressing SUD and trauma that are available have been mostly validated on males or specifically adapted for veteran populations. Mindfulness-Based Relapse Prevention (MBRP) is one evidence-based intervention that has demonstrated efficacy in reducing substance craving, relapse, and negative affect in a variety of SUD populations. It has also shown efficacy in incarcerated populations, ethnic minority women, and women offenders, all of which have higher levels of trauma exposure compared to normative samples. Research on Mindfulness-Based Interventions (MBIs) with trauma populations suggest that mindfulness skills can help decrease PTSD symptoms associated with avoidance and trauma-based cognitions, and that MBIs are not iatrogenic for trauma populations. A trauma informed adaptation of MBRP may thus offer an integrated intervention targeting both PTSD and SUD symptoms, and addressing the etiologies and maintaining factors underlying the comorbidity.

Given the particular needs and unique presentation of WST in substance use treatment settings, effective evidence-based interventions must be developed to improve treatment outcomes. The long-term goal of this line of research is to develop, examine and disseminate an adapted evidence-based treatment for comorbid SUD and PTSD for women survivors of trauma (WST). The primary objective of this study is to develop and evaluate an intervention that integrates trauma education and treatment approaches used in Cognitive Processing Therapy (CPT), an evidence-based intervention for PTSD, into the standard MBRP protocol to provide a trauma-informed approach to treating women in community-based substance use treatment settings. The development phase of the study will use focus groups with staff and clients from a women's residential treatment center who have completed the MBRP course to inform the integration of trauma education using the CPT manual into the MBRP protocol. Using a mixed-methods, pre-post, randomized-control design, WST (N=100) enrolled in a residential treatment program will be randomized by cluster into an experimental (TI-MBRP) or control (TAU) group to determine feasibility, acceptability, preliminary efficacy, and candidate mechanisms of TI-MBRP. To accomplish the primary objective, the following three aims are proposed:

Aim 1: Development and refinement of a Trauma Informed-Mindfulness Based Relapse Prevention (TI-MBRP) protocol. Informed by focus groups with staff and resident clients, a protocol integrating evidence-based practices for SUDs and PTSD will be developed for women in substance use treatment endorsing PTSD symptoms.

Aim 2: Determine feasibility and acceptability of TI-MBRP. Based on prior studies of MBRP in similar populations, we hypothesize TI-MBRP will be feasible and acceptable, as measured by recruitment and retention rates, weekly homework compliance, client participation in groups, and post-intervention client feedback.

Aim 3: Determine meaningful changes at pre-, post-, 1-, 3-, 6-, 9-, and 12-month follow-up assessment time points in SUD and trauma-related outcomes, and identify candidate mechanisms. We hypothesize that, as compared to TAU, participation in TI-MBRP will result in:

1. Significantly reduced trauma-related symptomology, craving, substance use, reactivity to negative affect, and experiential avoidance at post-intervention, and maintenance of treatment outcomes at 12-month follow-up.
2. Significant improvements in self-efficacy, coping skills, and mindfulness at post-intervention, and maintenance of treatment outcomes at 12-month follow-up.

Interested residents will be screened for eligibility based on the Inclusion/Exclusion Screening Tool, Breslau's Short Screening Scale, and Suicidal Behaviors Questionnaire. Eligible participants will be provided with a written informed consent. The PI will review the informed consent with participants and answer any questions or concerns that participants may have about study procedures, confidentiality, data analysis, and dissemination of results. Once written informed consent is obtained, participants will be notified of the group start date within one week of signing the consent form. Participants will be asked to complete a battery of paper-and-pencil assessments within one week prior to the start of the first session. Paper-and-pencil assessments will take no more than 60 minutes to complete.

Experimental and Treatment-As-Usual (TAU) groups will be implemented simultaneously for maximization of participants within the given time frame, totaling 10 groups over a 10-month period. Participants will complete a battery of self-report assessments at baseline. Then, using computer randomizing software, participants will be randomized by cluster into either an experimental or TAU group before the start of the first session. After the first session, all participants will be given an iPod touch with audio-recordings of guided meditation practices used in the intervention (i.e., body scan, breath awareness) to use as a part of their daily homework requirements. All iPod touch devices will include iMINDr, a software application developed to track frequency and duration of home meditation practice. Participants will then complete a post-course assessment battery within one week of the completion of the 4-week course. If participants are unable to be physically present to complete the post-course assessment, they will be offered a phone interview during which they will be administered self-report assessment measures orally.

One week after post-course assessment, participants will be invited to participate in an hour long, audio-recorded focus group to discuss helpful aspects of the intervention as well as what could be changed. Focus group audio recordings will be transcribed verbatim and analyzed in NVivo 11 by independent coders using a Constant Comparative Analysis.

Participants will be asked to complete additional paper-and-pencil assessments at 1-, 3-, 6-, 9-, and 12-months following post course. If participants are unable to physically attend follow-up assessment, they will be offered a phone interview with self-report assessments administered orally.

ELIGIBILITY:
Inclusion Criteria:

* 1) Be in the core learning phase of treatment at the Women's Residential Center (WRC)
* 2) Have a score of at least 4 on Breslau's Short Screening Scale for PTSD
* 3) Be age 18 to 70
* 4) Be fluent in speaking and reading English
* 5) Agree to randomization and attendance at treatment and assessment sessions
* 6) Be cleared for participation by appropriate clinic staff

Exclusion Criteria:

* 1) Report active suicidality as indicated by endorsing "Yes" to questions 5d - 5f in the Inclusion Exclusion Screening Form.
* 2) Endorse screening items indicating hallucinations or intense emotional lability
* 3) Have previously participated in an MBRP group in current or past treatment settings
* 4) Are in the stabilization or transition phase, versus core learning phase, of treatment
* 5) Fail to provide informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2020-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa C Somohano, MA, Principal Investigator — Pacific University
Locations (5):
- United States (5):
  - Beavterton Hazelden Betty Ford Foundation, Beaverton, Oregon
  - Lifeworks NW Walnut, Hillsboro, Oregon
  - Lifeworks NW Mountaindale, Mountaindale, Oregon
  - Springbrook Hazelden Betty Ford Foundation, Newberg, Oregon
  - Lifeworks NW Project Network, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Somohano VC, Kaplan J, Newman AG, O'Neil M, Lovejoy T. Formal mindfulness practice predicts reductions in PTSD symptom severity following a mindfulness-based intervention for women with co-occurring PTSD and substance use disorder. Addict Sci Clin Pract. 2022 Sep 16;17(1):51. doi: 10.1186/s13722-022-00333-2. PMID 36114577
- [Derived] Somohano VC, Bowen S. Trauma-Integrated Mindfulness-Based Relapse Prevention for Women with Comorbid Post-Traumatic Stress Disorder and Substance Use Disorder: A Cluster Randomized Controlled Feasibility and Acceptability Trial. J Integr Complement Med. 2022 Sep;28(9):729-738. doi: 10.1089/jicm.2021.0306. Epub 2022 May 31. PMID 35648046

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from community-based residential and intensive outpatient chemical dependency treatment centers in the Pacific Northwest. Facilities included three residential and two IOP clinics. Approximately 95% of women within these treatment facilities had a lifetime history of trauma, and approximately 88% were dually diagnosed with PTSD. Counselors and administrators assisted with recruitment via word of mouth, flyers, and announcements at weekly group meetings.
Pre-assignment Details: Participants who enrolled in the study agreed to complete an informed consent and screening procedure. Those who were eligible via our screening procedure completed baseline assessments prior to group assignment.
Groups:
- TI-MBRP: Trauma-Integrated Mindfulness-Based Relapse Prevention (TI-MBRP) will be a 4-week intervention integrating trauma intervention approaches based on Cognitive Processing Therapy (CPT), and gender-responsive interventions, into standard Mindfulness-Based Relapse Prevention (MBRP). TI-MBRP honors the spirit and cognitive-behavioral foundation of MBRP while introducing components of CPT. Each TI-MBRP session will include mindfulness practices that bring awareness to cognitive and behavioral processes of substance use, and how substance use may function as a mechanism to cope with trauma symptoms. Clients are trained to observe internal, triggering stimuli without reactively attempting to avoid these experiences through substance use as well as complete exercises that promote cognitive and emotional processing of traumatic events. Moreover, gender-focused themes will be discussed in relation to SUD and PTSD recovery such as parenting, interpersonal relationships, and empowerment.
Period: Overall Study
Arm/Group | TI-MBRP | Standard MBRP
Started | 38 | 45
Completed | 22 | 28
Not Completed | 16 | 17
Not completed — Lost to Follow-up | 7 | 11
Not completed — Withdrawal by Subject | 6 | 0
Not completed — Discharged from treatment | 3 | 6

BASELINE CHARACTERISTICS:
Population: The analysis population are women with comorbid PTSD and substance use disorder.
Groups:
- Total: Total of all reporting groups
Arm/Group | TI-MBRP | Standard MBRP | Total
Number analyzed (Participants) | 38 | 45 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.22 (10.28) | 32.55 (7.86) | 34.67 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 45 | 83
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 33 | 40 | 73
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 30 | 29 | 59
  More than one race | 1 | 5 | 6
  Unknown or Not Reported | 2 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 38 | 45 | 83

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: Number of participants who completed informed consent and screening, with at least 30% identifying as racial and/or ethnic minority.
Time Frame: Baseline
Population: Women in residential or intensive outpatient treatment substance use treatment from one of five clinics participating in the study during the time of study recruitment.
Measure: Count of Participants; unit: Participants
Groups:
- All Women Who Were Interested in Participation: All women who underwent informed consent and screening procedures.
Arm/Group | All Women Who Were Interested in Participation
Number analyzed (Participants) | 96
Participants | 96

2. Primary Outcome: Enrollment
Description: Percentage of eligible individuals who completed baseline measures.
Time Frame: Baseline
Population: Women with comorbid PTSD and substance use disorder.
Measure: Count of Participants; unit: Participants
Arm/Group | All Women Who Were Interested in Participation
Number analyzed (Participants) | 96
Participants | 83

3. Primary Outcome: Retention
Description: Percentage of participants who completed 1-month follow-up measures.
Time Frame: 8-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
Participants | 22 | 28

4. Primary Outcome: Trauma Symptoms by the Posttraumatic Checklist - Civilian (PCL-5) Scores
Description: 20-item screening instrument assessing PTSD symptoms. Each item is scored 0 - 4 (0 = Not at all, 1 = A little bit, 2 = Moderately, 3 = Quite a bit, 4 = Extremely). Total scores range from 0 - 80. Higher values indicate greater PTSD symptom severity.
Time Frame: Baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks, 36-weeks, 52-weeks
Population: Women with comorbid PTSD and Substance Use Disorder
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
score on a scale
  Baseline | 43.51 (15.28) | 48.55 (14.39)
  4-weeks | 35.41 (15.79) | 30.50 (13.86)
  8-weeks | 28.75 (14.98) | 21.82 (14.32)
  12-weeks | 30.17 (15.66) | 27.04 (16.50)
  24-weeks | 33.53 (18.50) | 29.84 (17.21)
  36-weeks | 27.67 (16.73) | 29.11 (14.72)
  52-weeks | 28.21 (21.01) | 28.69 (19.37)

5. Primary Outcome: Craving by the Penn Alcohol Craving Scale (PACS) Scores
Description: 5 items assessing frequency, intensity, and duration of alcohol or drug craving. Each item is scored 0-6 (0 = Never, 1 = Rarely , 2 = Occasionally , 3 = Sometimes, 4 = Often, 5 = Most of the time, 6 = Nearly all the time). Total scale scores range from 0 - 30. Higher scores indicate greater severity of alcohol and substance craving.
Time Frame: Baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks, 36-weeks, 52-weeks
Population: Women with PTSD and substance use disorder.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
score on a scale
  Baseline | 20.5 (7.76) | 21.31 (8.71)
  4-weeks | 8.33 (5.51) | 10.36 (8.48)
  8-weeks | 8.00 (5.03) | 6.86 (7.14)
  12-weeks | 7.38 (5.04) | 7.18 (6.61)
  24-weeks | 9.30 (7.41) | 5.15 (4.71)
  36-weeks | 8.67 (7.85) | 9.33 (7.61)
  52-weeks | 8.07 (6.19) | 9.15 (7.69)

6. Primary Outcome: Frequency of Alcohol and Substance Use by the NIDA Alcohol, Smoking, and Substance Involvement Test (ASSIST) Scores
Description: This self-report measure assesses frequency of alcohol and substance use, and misuse of prescription medication over the past 2 weeks, 30 days, and 3 months. Items are on a Likert scale, where 0 = "Not at all", 1 = "One or two days", 2 = "Several days", 3 = "More than half the days", and 4 = "Nearly every day". Total scare scores range from 0 - 44. Higher scores indicate greater frequency of use.
Time Frame: Baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks, 36-weeks, 52-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
score on a scale
  Baseline | .421 (1.26) | 1.15 (2.67)
  4-weeks | .454 (1.51) | .105 (.459)
  8-weeks | .333 (.707) | .000 (.000)
  12-weeks | .118 (.332) | .278 (1.18)
  24-weeks | 0.00 (0.00) | 0.00 (0.00)
  36-weeks | 2.36 (5.92) | .111 (.333)
  52-weeks | 4.14 (11.62) | .846 (2.51)

7. Secondary Outcome: Psychological Inflexibility and Experiential Avoidance by the Acceptance and Action Questionnaire - Substance Abuse (AAQ-SA) Scores
Description: 18-item self-report measure of experiential avoidance and psychological inflexibility related to substance abuse behaviors. Each item is scaled from 1 - 7, where 1 = "Never true", 2 = "Very seldom true", 3 = "Seldom true", 4 = "Sometimes true", 5 = "Frequently true", 6 = "Almost always true", and 7 = "Always true". Total scores range from 18 to 126. Higher scores indicate less psychological flexibility with regard to substance use.
Time Frame: Baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks, 36-weeks, 52-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
score on a scale
  Baseline | 84.13 (19.09) | 87.36 (18.43)
  4-weeks | 94.19 (15.64) | 100.37 (13.86)
  8-weeks | 97.77 (14.53) | 105.5 (13.49)
  12-weeks | 99.12 (16.07) | 107.86 (13.75)
  24-weeks | 89.69 (31.67) | 109.38 (12.45)
  36-weeks | 101.93 (21.35) | 110.22 (11.61)
  52-weeks | 103.79 (20.98) | 107.08 (13.35)

8. Secondary Outcome: Difficulties in Emotion Regulation Scale - Non-acceptance (DERS-NA)
Description: 36-item self-report measure of reaction to negative affect. This measure contains 6 subscales and a total score, and only the 6-item non-acceptance of emotion subscale (α = 0.85) was be used, which measures the degree to which an individual accepts their reaction to negative emotions. Items are scaled from 1 - 6, where 1 = "Almost never (1 - 10%)", 2 = "Sometimes (11 - 35%)", 3 = About half the time (36 - 65%)", 4 = "Most of the time (66 - 90%)", and 5 = "Almost always (91 - 99%)". Total subscale scores range from 6 to 30. Higher scores indicate less acceptance of negative affective states.
Time Frame: Baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks, 36-weeks, 52-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
score on a scale
  Baseline | 17.10 (5.59) | 17.55 (5.83)
  4-weeks | 14.66 (4.32) | 13.27 (5.04)
  8-weeks | 14.26 (6.73) | 11.77 (4.92)
  12-weeks | 14.62 (5.55) | 10.86 (5.55)
  24-weeks | 13.70 (5.06) | 10.92 (4.80)
  36-weeks | 13.07 (7.07) | 11.78 (5.33)
  52-weeks | 12.00 (5.52) | 11.53 (4.39)

9. Secondary Outcome: Five Facet Mindfulness Questionnaire - Short Form (FFMQ-SF)
Description: 24-item, self-report measure of mindfulness. The FFMQ-SF contains a total mindfulness score and 5 subscale scores measuring awareness, non-judgment, describing, observing, and non-reactivity. Items are scaled from 1 - 5, where 1 = "Never or very rarely true", 2 = "Rarely true", 3 = "Sometimes true", 4 = "Often true", and 5 = "Very often or always true". Subscale scores are combined to achieve a total score, which are presented in the data table below. Total scores range from 24 to 120. Higher scores indicate greater levels of mindfulness.
Time Frame: Baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks, 36-weeks, 52-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
score on a scale
  Baseline | 74.48 (11.85) | 72.71 (10.41)
  4-weeks | 78.19 (11.03) | 81.00 (12.65)
  8-weeks | 82.50 (8.87) | 88.10 (12.20)
  12-weeks | 80.29 (12.48) | 88.50 (14.49)
  24-weeks | 80.77 (12.13) | 93.69 (13.57)
  36-weeks | 88.53 (14.05) | 88.44 (12.96)
  52-weeks | 88.00 (12.27) | 91.38 (15.86)

10. Secondary Outcome: Coping Responses Inventory (CRI)
Description: The CRI is a self-report, 48-item questionnaire assessing coping resources in stressful situations, with subscales measuring approach-based coping and avoidant coping in difficult situations. Items are on a 4-point Likert scale varying from "Not at all" to "Fairly often". Subscale scores on approach- and avoidant-based coping range from 0 to 72, and each contain 24 items. Higher scores on the approach-based coping subscale indicates greater use of approach-based coping strategies when faced with a stressor. Higher scores on the avoidance-based coping subscale indicates greater use of avoidant-based coping strategies when faced with a stressor.
Time Frame: Baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks, 36-weeks, 52-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
score on a scale
  Baseline Avoidance | 15.72 (9.89) | 22.05 (14.07)
  Baseline Approach | 23.52 (15.58) | 28.77 (17.36)
  4-weeks Avoidance | 14.97 (8.64) | 16.51 (11.56)
  4-weeks Approach | 27.80 (10.89) | 31.27 (16.36)
  8-weeks Avoidance | 12.50 (9.50) | 15.03 (10.46)
  8-weeks Approach | 28.68 (13.70) | 33.14 (18.07)
  12-weeks Avoidance | 30.52 (11.01) | 28.41 (9.53)
  12-weeks Approach | 50.41 (9.51) | 48.57 (13.41)
  24-weeks Avoidance | 26.00 (8.40) | 23.85 (6.96)
  24-weeks Approach | 44.83 (13.66) | 50.54 (12.73)
  36-weeks Avoidance | 23.33 (6.98) | 22.67 (6.52)
  36-weeks Approach | 43.20 (13.43) | 46.22 (15.17)
  52-weeks Avoidance | 22.86 (9.20) | 30.54 (13.84)
  52-weeks Approach | 44.21 (12.04) | 50.84 (12.27)

11. Secondary Outcome: Drug Taking Confidence Questionnaire
Description: 8-item brief self-report questionnaire measuring confidence in avoiding, abstaining or moderating substance use across 8 categories of relapse precipitants. Items are scaled from 0 - 100 in increments of 20, where 0 = "Not confident at all" and 100 = "Very confident".
Time Frame: Baseline, 4-weeks, 8-weeks, 12-weeks, 24-weeks, 36-weeks, 52-weeks
Measure: Mean (Standard Deviation); unit: percentage of confidence in abstaining
Arm/Group | TI-MBRP | Standard MBRP
Number analyzed (Participants) | 38 | 45
percentage of confidence in abstaining
  Baseline | 43.36 (21.58) | 39.87 (27.33)
  4-weeks | 57.05 (19.12) | 61.22 (20.98)
  8-weeks | 55.97 (23.68) | 65.46 (19.37)
  12-weeks | 63.17 (15.75) | 63.23 (24.18)
  24-weeks | 55.60 (22.01) | 65.08 (20.80)
  36-weeks | 62.27 (21.93) | 72.00 (10.15)
  52-weeks | 62.14 (20.63) | 67.85 (12.59)

ADVERSE EVENTS:
Time Frame: Adverse event data were assessed through study completion, an average of 1 year, and collected quarterly (i.e., every three months).
Arm/Group | TI-MBRP | Standard MBRP
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/45
Other Adverse Events (participants affected / at risk) | 0/38 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT03505749/Prot_SAP_000.pdf